CLINICAL TRIAL: NCT00992485
Title: A Phase I Dose Escalation Clinical Study of ADIPOPLUS (Autologous Cultured Adipose-derived Stem Cell) for the Treatment of Crohn's Fistula to Evaluate Safety and Efficacy
Brief Title: Safety and Efficacy Study of Autologous Cultured Adipose -Derived Stem Cells for the Crohn's Fistula
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Anterogen Co., Ltd. (Industry)
Responsible Party: Mihyung Kim, Director
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANTG-ASC-201
Record Dates: First submitted 2009-09-29; First posted 2009-10-09 (Estimated); Last update posted 2010-05-10 (Estimated); Status verified 2010-05

CONDITIONS: Crohn's Fistula

ARMS (1):
- autologous adipose derived stem cell (Experimental)
  Interventions: Drug: ADIPOPLUS

INTERVENTIONS:
Drug: ADIPOPLUS — autologous adipose-derived stem cell

SUMMARY:
Up to date, a sure cure for Crohn's fistula has not known and the fistula recurrence rate is high. On 15 October 2008, orphan drug designation was granted by Korea FDA to Anterogen Co. Ltd., for human adipose-derived stem cell. In this study, patients are given injection of ADIPOPLUS in fistula site and followed for 8 weeks to test the safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Prior diagnosis of Crohn's disease
* patients who have Crohn's fistula
* negative for urine beta-HCG for woman of childbearing age
* agreement to participate, with signed informed-consent

Exclusion Criteria:

* patients who have allergy to bovine-derived materials or an anesthetic
* patients with a diagnosis of auto immune disease except for Crohn's disease
* Diagnosis of HBV, HCV, HIV and other infectious disease
* Patients who have a symptom of septicemia
* Patients with a diagnosis of active Tuberculosis
* Patients who are pregnant or breast-feeding
* Patients who are unwilling to use an "effective" method of contraception during the study
* Patients with a diagnosis of Inflammatory Bowel Disease except for Crohn's disease
* Patients who is sensitive to Fibrin glue
* Patients who have a clinically relevant history of abuse of alcohol or drugs
* Insufficient adipose tissue for manufacturing of ADIPOPLUS
* Patients who are considered not suitable for the study by investigator
* Patients who have history of surgery for malignant cancer in the past 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-11; Primary Completion 2009-09 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Efficacy: closure of fistula at week 8 Safety: - Clinically measured abnormality of laboratory tests and adverse events

SECONDARY OUTCOMES:
Closure of fistula | week 4
Investigator satisfaction | week 4 and week 8
Patient satisfaction | week 4 and week 8
Digital photography | day 1, week 4 and week 8

CONTACTS AND LOCATIONS:
Locations (1):
- Asan medical center, Seoul, South Korea